CLINICAL TRIAL: NCT01169194
Title: Multi-Center African-American Inflammatory Bowel Disease Study (MAAIS)
Acronym: MAAIS
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00041578; U01DK062431 (NIH)
Record Dates: First submitted 2010-06-16; First posted 2010-07-26 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; IBD; CD; UC; IC; African American IBD; African American CD; African American UC; African American IC; Black IBD; Black CD; Black UC; Black IC; African American Inflammatory Bowel Disease; African American Crohn's Disease; African American Ulcerative Colitis; African American Indeterminate Colitis; Black Inflammatory Bowel Disease; Black Crohn's Disease; Black Ulcerative Colitis; Black Indeterminate Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and derivatives from blood, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Affected: Patients with IBD
- Unaffected: Individuals who do not have IBD

SUMMARY:
The investigators are doing the research to discover genes that cause Inflammatory Bowel Disease (IBD) specifically in the African American population. African Americans with or without Crohn's disease or ulcerative colitis are eligible to join. If you agree to join the study, the investigators will ask for information about your health. The investigators will also ask you to give us a blood sample so that they may discover the genes that cause IBD. The blood sample may be collected at Johns Hopkins or any local facility convenient to you.

DETAILED DESCRIPTION:
This current protocol was established as part of an NIDDK initiative to further explore genetic factors associated with IBD. Specifically, the investigators are interested in identifying the genetic, environment and socio-economical components that contribute to the development of IBD in the African American population.

IBD is believed to be caused by a combination of environmental and genetic factors. Genetic data will be examined alongside potential environmental factors such as smoking, medications, environmental exposures, and some dietary factors. Since IBD is known to predominantly affect Western, industrialized areas of the world, the investigators will also inquire about participants' socioeconomic background in hopes of identifying any previously unknown factors in the AA population that may increase the risk of IBD. These potential environmental factors will be important in association analyses using covariates as these factors can obscure potential associations or interact with genetic factors and thus contribute to genetic associations. The investigators will also obtain information as to ancestry of parents and grandparents as to best match cases with unrelated controls of similar ancestry (e.g., Caribbean, recent European or recent African ancestry could cause genetic mismatch of a case and control). At the same time, the investigators will also collect similar information (smoking, medications, environmental exposures and dietary factors) from non-African Americans for the purpose of making direct comparisons for these parameters between the different racial groups to assess the contribution of non-genetic factors for susceptibility to the development of IBD.

This study calls for recruiting AA patients and ethnically matched controls (friend or spouse). These persons will provide us with a blood sample and with information requested on a questionnaire asking the following: clinical course and history of their IBD or their general health, smoking history, socioeconomic variables and specific dietary factors known in some populations to be related to IBD etiology. Access to medical records will be used to confirm diagnoses. The clinical characteristics of IBD obtained from medical records will be summarized in a phenotyping form using a standardized NIDDK IBDGC Phenotyping Operations Manual. Controls will be asked health history to identify potentially unrecognized IBD. DNA and other biospecimens will be purified from blood. Samples and data will also be shared with the NIDDK IBDGC for use in IBDGC research projects and will be processed and maintained at NIDDK repositories.

ELIGIBILITY:
Inclusion Criteria:

1. African Americans with a confirmed diagnosis of Inflammatory Bowel Disease (IBD)
2. African Americans without a diagnosis of IBD and without a family history of IBD for comparison purposes

Exclusion Criteria: Patients whose IBD cannot be confirmed

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with Inflammatory Bowel Disease
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2003-06 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
IBD Genes | Single visit, approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lazarev, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No